CLINICAL TRIAL: NCT02608528
Title: Serial [18F]Fluorodeoxyglucose ([18F]FDG )PET/CT as a Biomarker of Therapeutic Response in Anti-PD1/PDL1 Therapy
Status: Terminated | Type: Observational
Why Stopped: Poor Accrual
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 15515
Record Dates: First submitted 2015-11-17; First posted 2015-11-18 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: [18F]fluoroglucose(FDG)

SUMMARY:
Evaluation of FDG PET/CT to image immunotherapy response in adult thoracic cancer.

Compare pre- and post-treatment primary tumor uptake for FDG-PET/CT and correlate with clinical markers of response. PET/CT tumor metabolic response will also be correlated will to progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, at least 18 years of age
* Histologically confirmed non-small cell lung cancer or malignancy pleural mesothelioma with at least one site of disease > 1 cm by at least one type of standard imaging (e.g.

CT, chest x-ray, MRI)

* Recommended to start anti-PD1/PDL1 therapy.
* Obtaining pre-PD1/PDL1 therapy clinical re-staging [18F]FDG-PET/CT scan at the Hospital of the University of Pennsylvania.
* Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.
* Participants must be willing and able to comply with scheduled visits and imaging procedures in the opinion of the investigator or treating physician.

Exclusion Criteria

* Females who are pregnant or breast-feeding at the time of screening will not be eligible for this study. Female participants of child-bearing potential will have a urine pregnancy test at the time of the screening visit.
* Patients with only a single site of primary non-small cell lung cancer or malignancy pleural mesothelioma who have undergone or are recommended to undergo radiation therapy to that site will not be eligible, the inclusion of patients who may be undergoing radiation therapy to ancillary disease sites may be allowed to enter the study at the discretion of the PI if it is not felt to affect the ability to capture [18F]FDG information for at least one primary site of disease.
* Patients who have undergone cancer surgery removing a significant portion of active disease, in the opinion of an investigator, within 2 months prior to study enrollment will be excluded.
* Patients who have received prior immunotherapy.
* Patients with an active auto-immune disease (ie. Multiple sclerosis, rheumatoid arthritis, systemic lupus erythematosus, vasculitis).
* Inability to tolerate imaging procedures in the opinion of the investigator or treating physician
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator would compromise the subject's safety or successful participation in the study.
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women of any ethnicity with NSCLC deemed unresectable by CT or PET imaging criteria and planning to start anti-PD1/PDL1 therapy.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Number of inflammatory changes within the tumor | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sharyn Katz, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States